CLINICAL TRIAL: NCT03290911
Title: An Observational Retrospective Cohort Trial on Low Prognosis Infertile Patient's Accessing IVF Cycle Management
Brief Title: Retrospective Trial on Low Prognosis Infertile Patients
Status: Completed | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Collaborators: Merck Serono International SA (Industry)
Responsible Party: Sponsor
Other Study IDs: 15/17
Record Dates: First submitted 2017-09-19; First posted 2017-09-25 (Actual); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Infertility, Female; Fertility Disorders
Keywords: low responders
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main objective of this study is to analyze management of Controlled Ovarian Stimulation (COS) protocols in low prognosis patients, secondly to observe the clinical outcomes (Fertilization Rate, Pregnancy Rate, the Ongoing Pregnancy Rate and the Live birth Rate) and the total units of gonadotrophins consume per M2 oocyte retrieved in this subgroup.

DETAILED DESCRIPTION:
Humanitas Fertility Center maintains an external audit anonymized electronic research queries system, exported from a certified only access web database, which at time of this analysis (cycles at December 31th 2016) include 26,883 consecutive fresh non-donors IVF cycles. Patients who underwent these cycles had consented in writing that their medical records could be used for research purposes, as long as the patients' anonymity was protected and confidentiality of the medical record was assured. Since both of these conditions were met, this study has been approved on March 2th 2017 with an expedited review and approval protocol by the center's Institutional Review Board (IRB).

At least 2,000 expected low prognosis patients in the Humanitas Fertility Center Database out of 12,545 cycles performed in the period 2010-2015 with completed pregnancy follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age ≤ 44
* Body Mass Index; 18 ≤ BMI ≥ 27
* Number of oocytes retrieved ≤ 9
* Cycles performed between January 2010 - December 2015

Exclusion Criteria:

* Age > 44
* Number of oocytes retrieved ≥ 10
* Abnormal uterine cavity
* Endometriosis III-IV stage or adenomyosis
* Testicular spermatozoa PGS (Preimplantation Genetic Screening) cycles

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: 26,883 consecutive fresh non-donors IVF cycles. Patients who underwent these cycles had consented in writing that their medical records could be used for research purposes, as long as the patients' anonymity was protected and confidentiality of the medical record was assured. Since both of these conditions were met, this study has been approved on March 2th 2017 with an expedited review and approval protocol by the center's Institutional Review Board (IRB).
  At least 2,000 expected low prognosis patients in the Humanitas Fertility Center Database out of 12,545 cycles performed in the period 2010-2015 with completed pregnancy follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 26883 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
induction protocol type | 6 years
  number of antagonist and agonist protocols/ total numbers

SECONDARY OUTCOMES:
Fertilization Rate | 6 years
  fertilized oocytes/ number of oocytes used
Pregnancy Rate | 6 years
  number of gestational sacs/ number of embryos transferred
Ongoing Pregnancy Rate | 6 years
  number of pregnancy > 20 weeks/ total pregnancies
Live Birth Rate | 6 years
  number babies born/ total pregnancies

REFERENCES:
- [Derived] Levi-Setti PE, Zerbetto I, Baggiani A, Zannoni E, Sacchi L, Smeraldi A, Morenghi E, De Cesare R, Drovanti A, Santi D. An Observational Retrospective Cohort Trial on 4,828 IVF Cycles Evaluating Different Low Prognosis Patients Following the POSEIDON Criteria. Front Endocrinol (Lausanne). 2019 May 8;10:282. doi: 10.3389/fendo.2019.00282. eCollection 2019. PMID 31139146